CLINICAL TRIAL: NCT00512213
Title: Immunonutrition Versus Standard Enteral Nutrition Before Major Surgery: A Single-center Double-blinded Controlled Randomized Superiority Trial
Brief Title: Immunonutrition Versus Standard Enteral Nutrition Before Major Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, professor of surgery, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P00/07 CHV
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Major Abdominal Surgery
Keywords: preoperative Immunonutrition; major abdominal surgery; complication
MeSH Terms: interventions — Immunonutrition Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Immunonutrition containing RNA, omega-3-FAs, arginine
  Interventions: Dietary Supplement: Immunonutrition for 5 days preoperative
- 2 (Active Comparator): Standard enteral nutrition: isocaloric and isonitrogeneous but w/o active ingredients
  Interventions: Dietary Supplement: Standard enteral nutrition for 5 days preoperative

INTERVENTIONS:
Dietary Supplement: Immunonutrition for 5 days preoperative — Impact vs Meritene
  Other Names: Impact, Meritene
  Arms: 1
Dietary Supplement: Standard enteral nutrition for 5 days preoperative — Impact vs Meritene
  Other Names: Impact vs Meritene
  Arms: 2

SUMMARY:
The aim of this trial is to compare preoperative Imunnonutrition with standard enteral nutrition regarding morbidity after major abdominal surgery in patients with NRS greater 3.

The primary end point is the complication rate until 30 days after surgery.

DETAILED DESCRIPTION:
Malnutrition affects about 20-50% of all patients in hospital [1, 2]. Major surgery further increases postoperative malnutrition and immunity reduction. Therefore, postoperative complication and infection rates after major surgery exceed 30% [3-6].

The nutritional risk score (NRS) [1] is based on the ESPEN (European society of parenteral and enteral nutrition) screening guidelines and identifies patients who are likely to benefit from nutritional support. Patients with a NRS ≥ 3 are considered severely undernourished, or to have a certain degree of severity of disease in combination with certain degree of malnutrition [7].

In a prospective cohort study patients with a NRS ³ 3 had significant more infectious and overall complications after major abdominal surgery [4, 7, 8]. Several studies showed a benefit by nutritional support on complications [3, 5, 6]. International guidelines suggest therefore preoperative oral nutritional support for malnourished patients undergoing major surgery [9]. However, it remains controversial whether standard enteral nutrition (SEN) or immunonutrition (IN) is preferable [9].

IN, containing arginine, ribonucleic acid and omega-3 polyunsaturated fatty acids aims to improve the nutritional status, immunological function and clinical outcome [5, 10].

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted for elective major abdominal surgery:

  * Open and laparoscopic esophageal, gastric, hepatic, pancreatic, intestinal and colorectal surgery and with a NRS ≥ 3.

Exclusion Criteria:

* Age < 18 years
* No informed consent
* Emergency situation
* Patients not speaking french or german.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
complications after surgery | 30 days

SECONDARY OUTCOMES:
hospital stay, patient compliance, Interleukin-6 and 10 plasma level | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Demartines, MD, Study Chair — Department of Visceral Surgery, University Hospital Center, Lausanne, Switzerland
Locations (1):
- Department of Visceral Surgery, University Hospital Center, Lausanne, Switzerland